CLINICAL TRIAL: NCT05537623
Title: Preventing Suicide With Safe Alternatives for Teens and Youths (SAFETY) - A Randomized Controlled Feasibility Trial
Brief Title: Preventing Suicide With Safe Alternatives for Teens and Youths (SAFETY)
Acronym: SAFETYF2022
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Johan Bjureberg, Associate Professor, Region Stockholm
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAFETY
Record Dates: First submitted 2022-08-10; First posted 2022-09-13 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Suicide and Self-harm
MeSH Terms: conditions — Suicide; Self-Injurious Behavior | interventions — Safety; Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Safe Alternatives for Teens and Youths (SAFETY) (Experimental): SAFETY is a transdiagnostic cognitive-behavioral family treatment informed by Dialectical Behavior Therapy (DBT) and Multisystemic Therapy (MST). The twelve week long treatment is principle based, structured in phases, and individually tailored based on a cognitive-behavioral fit analysis that specifies key risk and protective processes. Each session contains one individual component for youth and parents respectively, and one family component where youth and parents work together with therapists to practice skills identified as critical for preventing future suicidal behavior. Treatment targets are arranged in a SAFETY Pyramid, consisting of (a) safe settings; (b) safe people; (c) safe activities and actions; (d) safe thought; and (e) safe stress reactions, emphasizing strengthening protective support and validation within the family and/or social environment surrounding the youth.
  Interventions: Behavioral: Safe Alternatives for Teens and Youths (SAFETY)
- Supportive Therapy (Active Comparator): Supportive Therapy is a manualized client-centered therapy. The Supportive Therapy will be adapted to match SAFETY to control for nonspecific treatment factors such as therapist characteristics, time, and treatment exposure. The Supportive Therapy program consists of twelve weekly individual sessions with the youth, focusing on the therapeutic supporting relationship between the therapist and the youth, and follow-ups with parents. Therapeutic strategies include acceptance and validation, to increase feelings of connectedness and belonging and counteract thwarted belongingness, helplessness, and hopelessness. Cognitive-behavioral techniques (e.g., active modeling, problem-solving training, cognitive restructuring) are not allowed.
  Interventions: Behavioral: Supportive Therapy

INTERVENTIONS:
Behavioral: Safe Alternatives for Teens and Youths (SAFETY) — Please see description of experimental arm (arm one)
  Arms: Safe Alternatives for Teens and Youths (SAFETY)
Behavioral: Supportive Therapy — Please see description of active comparator arm (arm two)
  Arms: Supportive Therapy

SUMMARY:
Suicide is the leading cause of death in the age span 10-19 years in Sweden. The most robust predictor of future suicide attempt and suicide death is prior suicide attempt. Yet, most youths presenting with suicidal behavior to the Child and Adolescent Mental Health Services (CAMHS) in Stockholm, Sweden are not offered evidence-based care directly targeting suicide risk. Safe Alternatives for Teens and Youths (SAFETY) is a novel scalable suicide prevention program designed to fill this critical gap. SAFETY is a cognitive behavioral family treatment incorporating elements from Dialectical Behavior Therapy and Multisystemic Therapy. SAFETY has shown promise in reducing suicide attempts in two small-N trials. In a randomized controlled feasibility trial, the investigators will examine the feasibility of SAFETY and an active control condition named Supportive Therapy at post-treatment, 3 and 12 months after treatment on youth suicidal behavior. Evaluations of feasibility, acceptability, and safety based on data from this pilot trial will guide and inform the design of a full-scale randomized controlled trial.

DETAILED DESCRIPTION:
Research questions:

1. Is it feasible (operationalized as participation in treatment, completed homework assignments, reported adverse events) to offer SAFETY to youths with suicidal behavior and their caregivers within the CAMHS?
2. Is it feasible (operationalized as participation in treatment, completed homework assignments, reported adverse events) to offer Supportive Therapy as an active control treatment to youths with suicidal behavior and their caregivers within the CAMHS?
3. Is the planned procedure and design (recruitment, blinded assessors, randomization and data attrition) of the study feasible?
4. What are the proportions of suicidal behavior in the group randomized to SAFETY group and the group randomized to Supportive Therapy, respectively?
5. Is participation in SAFETY and Supportive Therapy associated with improved emotion regulation, perceived social support, and family function, and how large are the effects (suggested treatment processes)?
6. Is participation in SAFETY and Supportive Therapy associated with improvements in nonsuicidal self-injury, depression, anxiety, and other outcomes, and how large are the effects (outcomes)?
7. How do the youths and caregivers experience participation in SAFETY and Supportive Therapy, respectively?

ELIGIBILITY:
Inclusion Criteria:

* Suicidal behavior (defined as suicide attempt, interrupted suicide attempt, aborted suicide attempt, or preparatory behavior) in the last 3 months
* Age 10-17 years
* At least one primary caregiver willing to participate in treatment

Exclusion Criteria:

* Symptoms requiring other immediate treatment (e.g. psychosis, severe anorexia nervosa)
* Ongoing treatment with DBT
* Individual or life circumstances that could complicate or make treatment participation impossible, or that require immediate intervention (e.g., violence in close relationships; intellectual disability)
* Insufficient understanding of the Swedish language

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Number of completed assessments at week 12 | week 12
  Defined as number of completed assessments at end of intervention (week 12)
Number of completed assessments at 3 months follow-up | 3 months follow-up
  Defined as number of completed assessments 3 months after end of intervention
Number of completed assessments at 12 months follow-up | 12 months follow-up
  Defined as number of completed assessments 12 months after end of intervention
The fraction of eligible participants who consent to inclusion and randomization | week 12
  The fraction of potential participants will be determined as the number of eligible persons compared to the number of randomized persons.
Compliance | week 12
  Compliance will be defined as number of completed sessions.
Credibility/Expectancy Scale (CEQ) | week 1 (youth and parent reported)
  The CEQ is a 6-item measure of treatment credibility and expectancy. Scale points ranges from 0-9 and 0-100%, where a higher score indicates a better outcome.
Client Satisfaction Questionnaire (CSQ) | week 12 (youth and parent reported)
  The CSQ-8 is an 8-item self-rated 4-point scale, measuring different aspects of satisfaction with treatment, e.g. perception of quality of treatment, if the treatment adequately addressed their needs and overall satisfaction. Total range is 8 to 32, with higher values indicating higher satisfaction. Mean in total satisfaction scores on the CSQ-8 for each treatment group at end of treatment will be reported.
Adverse events | week 12 (youth and parent reported)
  Participants are asked to report and rate the discomfort of the eventual adverse events caused by their participation in the treatment.
Columbia Suicide Severity Rating Scale (C-SSRS) as exploratory clinical outcome | week 0 (clinician reported)
  The C-SSRS is a 22-item measure assessing the frequency and severity of suicidal ideation, suicidal behaviors, and self-harm. The C-SSRS will be administered as a clinical interview at baseline (week 0).
Columbia Suicide Severity Rating Scale (C-SSRS) as exploratory clinical outcome | once every week during treatment (week 1-11 after baseline; youth reported)
  See description above (outcome 9). The C-SSRS will be administered as a self-rated measure for weekly assessments during treatment.
Columbia Suicide Severity Rating Scale (C-SSRS) as exploratory clinical outcome | week 12 (end of treatment; clinician reported)
  See description above (outcome 9), The C-SSRS will be administered as a clinical interview.
Columbia Suicide Severity Rating Scale (C-SSRS) as exploratory clinical outcome | 3 months after end of treatment (clinician reported)
  See description above (outcome 9), The C-SSRS will be administered as a clinical interview.
Columbia Suicide Severity Rating Scale (C-SSRS) as exploratory clinical outcome | 12 months after end of treatment (clinician reported)
  See description above (outcome 9), The C-SSRS will be administered as a clinical interview.

SECONDARY OUTCOMES:
Difficulties In Emotion Regulation Scale (DERS) | Change from baseline, week 12 (end of treatment), 3 months and 12 months after end of treatment (youth and parent reported)
  The DERS is a measure of difficulties in emotion regulation, with 36 items rated on a 1-5 Likert scale, with a higher score indicating greater difficulties with emotion regulation.
Brief 16-item Version of the Difficulties In Emotion Regulation Scale (DERS-16) | Change from baseline, once every week during treatment (week 1-11; youth reported)
  DERS-16 is a brief 16-item version of the DERS, see description above, with 16 items rated on a 1-5 Likert scale, with a higher score indicating greater difficulties with emotion regulation.
Cognitive Emotion Regulation Questionnaire (CERQ) | Change from baseline, week 12 (end of treatment), 3 months and 12 months after end of treatment (youth reported)
  The CERQ is a measure of cognitive emotion regulation, with 36 items on a Likert scale ranging from 1-5. A higher score indicates greater difficulties with cognitive emotion regulation.
Behavioral Emotion Regulation Questionnaire (BERQ) | Change from baseline, week 12 (end of treatment), 3 months and 12 months after end of treatment (youth reported)
  The BERQ is a measure of behavioral emotion regulation, with 20 items on a Likert scale ranging from 1-5. A higher score indicates greater difficulties with behavioral emotion regulation.
Emotion Beliefs Questionnaire (EBQ) | Change from baseline, week 12 (end of treatment), 3 months and 12 months after end of treatment (youth reported)
  The EBQ is a measure of emotion beliefs, with 16 items on a Likert scale ranging from 1-7. A higher score indicates more maladaptive beliefs about emotions.
Perth Alexithymia Questionnaire (PAQ) | Change from baseline, week 12 (end of treatment), 3 months and 12 months after end of treatment (youth reported)
  The PAQ is a measure of how emotions are perceived and experienced, with 24 items on a Likert scale ranging from 1-7. A higher score indicates greater difficulties related to alexithymia.
Multidimensional Scale of Perceived Social Support (MSPSS) | Change from baseline, once every week during treatment (week 1-11), week 12 (end of treatment), 3 months and 12 months after end of treatment (youth reported)
  The MSPSS is a measure of perceived social support, with 12 items on a Likert scale ranging from 1-7. A higher score indicates higher level of perceived social support.
Systemic Clinical Outcome and Routine Evaluation, 15 item version (SCORE-15) | Change from baseline, once every week during treatment (week 1-11), week 12 (end of treatment), 3 months and 12 months after end of treatment (youth reported)
  The SCORE-15 is a measure of family function, with 15 items on a Likert scale ranging from 1-5. A higher score indicates greater family function.
Deliberate Self-Harm Inventory - Youth version (DSHI-Y) | Change from baseline, once every week during treatment (week 1-11), week 12 (end of treatment), 3 months and 12 months after end of treatment (youth reported)
  The DSHI-Y is a 7-item measure assessing occurrence, method, frequency of deliberate self-harm. A higher score indicates higher frequency and severity of self-harm. The DSHI-Y will be administered as a clinical interview at baseline, post and follow-up, and as a self-rated measure for weekly assessments.
Revised Children's Anxiety and Depression Scale, short (RCADS-S) | Change from baseline, week 12 (end of treatment), 3 months and 12 months after end of treatment (youth reported)
  The RCADS-S, a shortened version of the Spence Child Anxiety Scale, is a child self-report measure of anxiety- and depression-related psychopathology. Total range is 0-45, Likert scale ranging from 0-3, with higher values representing a worse outcome.
Beck's Hopelessness Scale (BHS) | Change from baseline, week 12 (end of treatment), 3 months and 12 months after end of treatment (youth and parent reported)
  The BHS is a measure of hopelessness, with 20 dichotomous "true/false" items. A higher score indicates greater difficulties related to hopelessness.
1-item version of the Perceived Criticism Measure (PCM - 1 item version) | Change from baseline, week 12 (end of treatment), 3 months and 12 months after end of treatment (youth reported)
  The PCM - 1 item version is a measure of expressed emotion, consisting of one question on a Likert scale ranging from 0-10, about how critical an emotionally important individual is perceived to be by the rater.
Borderline Symptom List Supplement (BSL-Supplement) | Change from baseline, once every week during treatment (week 1-11), week 12 (end of treatment), 3 months and 12 months after end of treatment (youth reported)
  The BSL-Supplement is a 11-item measure of self-destructive behaviors. Higher score indicates higher frequency of self-destructive behaviors.
Dialectical Behavior Therapy - Ways of Coping Checklist (DBT-WCCL) | Change from baseline, week 12 (end of treatment), 3 months and 12 months after end of treatment (youth reported)
  The DBT-WCCL is a measure of use of DBT skills use and dysfunctional ways of coping with emotions. Higher average score in the skills use subscale and lower average scores in the dysfunctional coping subscales indicate greater functional coping.
CRAFFT | Change from baseline, week 12 (end of treatment), 3 months and 12 months after end of treatment (youth reported)
  CRAFFT is a 9-item screening measure of alcohol and substance use. A higher score indicates greater difficulties related to substance use.
Pittsburgh Sleep Quality Index (PSQI) | Change from baseline, week 12 (end of treatment), 3 months and 12 months after end of treatment (youth reported)
  The PSQI is a 18-item measure of sleep problems. A higher score indicates greater sleep problems.
The Coping with Children's Negative Emotions Scale - Adolescent Version (CCNES-A) | Change from baseline, week 12 (end of treatment), 3 months and 12 months after end of treatment (parent reported)
  The CCNES-A is a measure of parental coping responses in response to adolescents' negative emotions. The CCNES-A version used in this trial consists of nine hypothetical scenarios accompanied by six types of responses, rated on a Likert scale ranging from 1-7.
Patient Health Questionnaire-9 (PHQ-9) | Change from baseline, week 12 (end of treatment), 3 months and 12 months after end of treatment (parent reported)
  The PHQ-9 is a measure of depression, with 10 items on a Likert scale ranging from 0-3. Higher score indicates greater depressive symptoms.
Generalized anxiety disorder 7-item scale (GAD-7) | Change from baseline, week 12 (end of treatment), 3 months and 12 months after end of treatment (parent reported)
  The GAD-7 is a measure of anxiety, with 7 items on a Likert scale ranging from 0-3. Higher score indicates greater anxiety symptoms.
The Work and Social Adjustment Scale, youth version (WSAS-Y) - adolescent and parent versions | Change from baseline, week 12 (end of treatment), 3 months and 12 months after end of treatment (youth and parent reported)
  WSAS-Y is a measure of impaired functioning in school, everyday life, friends and social life, recreation and hobbies and family and close relationships. The scale generates a global score ranging from 0 to 40, with higher scores indicating greater impairment.
Trimbos/iMTA questionnaire for Costs associated with Psychiatric illness (TIC-P) | Change from baseline, week 12 (end of treatment), 3 months and 12 months after end of treatment (parent reported)
  The TIC-P is a 37 item measure assessing healthcare and societal resource use, including for example items on healthcare resource use, medications, school absenteeism, and parental productivity loss. In the present trial no health economic evaluations will be conducted. Rather this instrument is included to gain feasibility data in preparation of a planned larger randomized controlled trial. Therefore, no data on TiC-P will be reported in this trial.
Child Health Utility 9D (CHU-9D) | Change from baseline, week 12 (end of treatment), 3 months and 12 months after end of treatment (youth reported)
  The CHU-9D is a measure of health related quality of life, with 9 items on a Likert scale ranging from 1-5. A higher score indicates greater health-related quality of life.
Children's Global Assessment Scale (CGAS) | Change from baseline, week 12 (end of treatment), 3 months and 12 months after end of treatment (clinician reported)
  The CGAS is a single item clinician rated 1-100 scale that integrates psychological, social, and academic functioning in children as a measure of psychiatric disturbance. Higher values represent a better outcome.
The Clinical Global Impressions -Severity and Improvement scales (CGI-S; CGI-I) | Change from baseline, week 12 (end of treatment), 3 months and 12 months after end of treatment (clinician reported)
  The CGI-S and CGI-I are clinician rated 1-item scales ranging from 1-7 where higher ratings indicate greater symptom severity (CGI-S), and greater symptom improvement (CGI-I), respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Bjureberg, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Stockholm Regional Council, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karemyr M, Bellander M, Ponten M, Ohlis A, Flygare O, Wallden Y, Kuja-Halkola R, Hadlaczky G, Mataix-Cols D, Asarnow JR, Hellner C, Hughes JL, Bjureberg J. Preventing suicide with Safe Alternatives for Teens and Youths (SAFETY): a randomised feasibility trial. BMJ Ment Health. 2025 Apr 29;28(1):e301575. doi: 10.1136/bmjment-2025-301575. PMID 40306939